CLINICAL TRIAL: NCT01595087
Title: A Phase I/II Study of ODX (Osteodex) in Metastatic Castration Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DexTech Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODX-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Prostate Cancer Metastatic
Keywords: CRPC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Osteodex, infusion (Experimental): Osteodex
  Interventions: Drug: Osteodex

INTERVENTIONS:
Drug: Osteodex — Seven cohorts; Dose cohort 1; 0.1 mg/kg given every third week, maximum 7 times. Dose cohort 2; 0.3 mg/kg given every third week, maximum 7 times. Dose cohort 3; 0.6 mg/kg given every third week, maximum 7 times. Dose cohort 4; 0.9 mg/kg given every third week, maximum 7 times. Dose cohort 5; 1.2 mg/kg given every third week, maximum 7 times. Dose cohort 6; 1.5 mg/kg given every third week, maximum 7 times. Dose cohort 7; 3.0 mg/kg given every third week, maximum 7 times.
  Other Names: Castration resistant prostate cancer

SUMMARY:
This phase I/IIa study is a multi-center, prospective, open-label study evaluating safety and biological efficacy of up to six dose levels of Osteodex of patients with metastatic castration resistant prostate cancer (CRPC). Osteodex is a poly-bisphosphonate containing three known substances; dextran, alendronate and guanidine.

The objective of the study is to define the maximum tolerable dose of Osteodex when given every third week. The following objectives will also be evaluated: overall survival, PSA response, response markers related to bone metabolism (S-ALP and U-NTx), Quality of Life and assessment of pharmacokinetic parameters.

DETAILED DESCRIPTION:
Males, diagnosed with CRPC, who fulfil the inclusion criteria and does not have any exclusion criteria, will be asked to participate in the study. The subject will be informed orally and in writing about the study procedures and give written informed consent, prior to study start. At the screening visit the following examinations are performed: Physical examination, medical history and concomitant medication. Heart rate, blood pressure, weight, body temperature and respiratory rate are measured. Blood samples are drawn and urine sample is collected. ECG is performed. At the next visit, baseline, the subject is examined physically and heart rate, blood pressure, weight, body temperature and respiratory rate are measured, ECG is performed, blood samples drawn and urine sample collected. FACT-P questionnaire is filled out by the subject. Adverse events and concomitant medication is documented and the first dose of the investigational product is given. The subject will be consecutively assigned to the dose cohorts, starting with the lowest dose cohort, cohort one out of seven cohorts.

Then the subject is surveyed during 24 hours at the hospital. Prior to discharge from the hospital the same examinations are done as described above.

The duration of the study for the individual subject will be approximately 25 weeks from screening to the follow-up visit 3 weeks after the last dose. Each subject will receive at least 4 doses and maximum 7 doses of investigational product.

A Data Monitoring Committee (DMC) will be designated and will be responsible to monitor/review all study related safety data. After review of safety data the DMC will provide recommendation as to whether the dose escalation can proceed as planned according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent form.
* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate.
* Failing or not tolerating docetaxel therapy or for other reasons not suitable for such therapy.
* Evidence of metastatic disease from bone scan (bone lesions) or other imaging modality.
* Evidence of PSA progression in two consecutive determinations at minimum 1 week interval
* Castrate levels of serum testosterone ≤1.7 nmol/L.
* Performance status ECOG 0-2
* Laboratory requirements:
* Haematology:
* Neutrophils ≥ 1.5 x 109/l
* Haemoglobin ≥ 90 g/l
* Platelets ≥ 100 x 109/l

Hepatic function:

* Total S-bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* AST (SGOT) / ALT (SGPT) ≤ 2.5 times ULN

Renal function:

* S-Cr ≤ 1.5 times the upper limit of normal (ULN)

Electrolytes:

* S-sodium, S-potassium, S-calcium (S-albumin corrected), S-phosphate, S-magnesium, all within normal ranges.
* No evidence (≤5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin)
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Concurrent use of other anti-cancer agents or treatments, with the following exception: a stable dose of LHRH agonist/antagonist, polyestradiol phosphate, bicalutamide, flutamide or cyproterone is allowed.
* Any treatment modalities involving chemotherapy, radiation or major surgery within 4 weeks prior to treatment in this study.
* Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to start of study treatment.
* Any condition, including the presence of laboratory abnormalities, which confounds the ability to interpret data from the study or places the patient at unacceptable risk if he participates in the study.
* Known brain metastases.
* Dental surgery (dental extraction), periodontal disease, local trauma including poorly fitting dentures within 6 months prior to the first dose of study drug.
* Treatment with bisphosphonates within 4 weeks prior to first dose of study medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerable dose (MTD) of Osteodex. | up to 21 weeks
  The MTD will be defined as the dose that is a predecessor to the dose where dose limiting toxicity (DLT, e.g., lack of recovery to baseline of serum creatinine (S-Cr), clinically significant abnormalities in test results for haematology, liver function, electrolytes, calcium, clinically significant ECG changes) occurs within 3 weeks after administration for at least 1 among 4 subjects. In case such dose limiting toxicity (DLT) is not observed for any doses the maximum dose at 1.5 mg/kg will be defined as the MTD.

SECONDARY OUTCOMES:
Evaluation of overall survival | Baseline and 21 weeks
PSA response | Baseline and 21 weeks
Response markers related to bone metabolism (S-ALP and U-NTx) | Baseline and 21 weeks
Quality of Life | Baseline and 21 weeks
  FACT-P questionnaire
Assessment of blood half life | pre-infusion and 30 min, 1 hr, 2 hrs, 3 hrs and 6 hrs post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Anders R Holmberg, CEO, Study Director — DexTech Medical AB
Locations (3):
- Sweden (3):
  - Oncology clinic, Skånes Universitetssjukhus i Lund, Lund, Lund
  - Urology clinic, Södersjukhuset AB, Stockholm, Stockholm County
  - Oncology clinic, Norrlands Universitetssjukhus, Umeå, Umeå